CLINICAL TRIAL: NCT01519232
Title: A Pilot Study of Changes in Hepatic Function During Radiation Therapy Using Hepatobiliary SPECT
Brief Title: A Study of Changes in Hepatic Function During Radiation Therapy Using Hepatobiliary Single Photon Emission Tomography (SPECT)
Status: Completed | Type: Observational
Sponsor: University of Michigan Rogel Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: UMCC 2007-110; HUM00015656 (Other: University of Michigan Medical IRB)
Record Dates: First submitted 2011-09-23; First posted 2012-01-26 (Estimated); Last update posted 2015-05-18 (Estimated); Status verified 2015-05

CONDITIONS: Hepatocellular Carcinoma
Keywords: hepatocellular carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Liver Irradiation: patients already scheduled to undergo liver irradiation
  Interventions: Radiation: Liver Irradiation

INTERVENTIONS:
Radiation: Liver Irradiation — Patients already scheduled to undergo radiation treatment

SUMMARY:
Radiation-induced liver disease (RILD) is a syndrome characterized by the development of anicteric ascites approximately 2 weeks to 4 months after hepatic irradiation. Previous studies have shown that both the volume of liver irradiated and the dose of radiation delivered are prominent factors for development of RILD. While use of a population-based normal tissue complication probability model allows investigators to limit the risk of RILD to a clinically acceptable level, a test that permits investigators to determine an individual's risk of RILD during the course of treatment may allow for individualized treatment modifications, either to prevent toxicity or increase efficacy.

DETAILED DESCRIPTION:
Early, but subclinical physiologic changes in the liver may be associated with the future development of RILD. There are currently limited data on how a local change in hepatic function associates with regional radiation dose, and how the change of hepatic function during and after radiation therapy (RT) associates with RILD. In the present study, a radiological methodology that is minimally invasive will be used to measure volumetric hepatic functions in patients with intrahepatic malignancies before, during, and after a course of fractioned radiation therapy.

ELIGIBILITY:
Inclusion Criteria:

* cancer patients undergoing radiation of the Liver
* women and men who agree to avoid pregnancy
* life expectancy of at least 6 months

Exclusion Criteria:

* pregnant women
* breatsfeeding women
* prisoners

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: cancer patients undergoing radiation of the Liver
Sampling Method: Probability Sample
Enrollment: 23 (Actual)
Dates: Start 2008-08; Primary Completion 2012-06 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Changes in hepatobiliary single photon emission tomography (SPECT) after radiation therapy | 6 months
  Changes in SPECT, which reflect hepatocyte function, will be correlated with specific regions of radiation dose to determine a relationship between dose and radiation-induced damage.

SECONDARY OUTCOMES:
measuring values between regional radiation dose and local hepatic function as measured by hepatobiliary SPECT, in normal liver parenchyma | 6 months
  dynamic hepatobiliary single photon emission tomography (SPECT) values will assess changes in hepatocyte function in patients with intrahepatic malignancies receiving radiation therapy. Perhaps a relationship between SPECT and dosage can be determined.

CONTACTS AND LOCATIONS:
Overall Officials: Mary Feng, MD, Principal Investigator — University of Michigan Rogel Cancer Center
Locations (1):
- University of Michigan Comprehensive Cancer Center, Ann Arbor, Michigan, United States